CLINICAL TRIAL: NCT02431377
Title: Acceptability and GI Tolerance of an Alpha-lactalbumin-enriched Formula: An Uncontrolled, Open-label, Descriptive Study
Brief Title: Acceptability and GI Tolerance of an Alpha-lactalbumin-enriched Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 14.23.INF
Record Dates: First submitted 2015-04-07; First posted 2015-05-01 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-10

CONDITIONS: Infant Formula Intolerance
Keywords: infant formula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- S-26 Gold (Experimental): Standard Infant Formula containing enriched with alpha-lactalbumin
  Interventions: Other: S-26 Gold

INTERVENTIONS:
Other: S-26 Gold — A commercial whey protein dominant, first age formula, containing whey protein concentrate with alpha-lactalbumin

SUMMARY:
A single center, non-controlled trial to document the gastrointestinal (GI) tolerability of the study formula (SF), containing a whey protein concentrate enriched with alpha-lactalbumin (WPC alpha-lac) fed for 6 weeks to healthy, term infants.

DETAILED DESCRIPTION:
The purpose of this study is to examine the tolerable and acceptability of an infant formula with with a Whey protein concentrate containing alpha-lactalbumin as measure by GI tolerance, and eating behaviors.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Healthy, full term, singleton infant
3. Be between 28±7 days post-natal age
4. Infants at enrollment, weight-for-age ≥ 5th and ≤ 95th percentile according to World Health Organization growth tables / charts
5. Infants must be exclusively consuming and tolerating a cow's milk infant formula for a minimum of 3 consecutive days and parent(s)/LAR must have previously made the decision to continue to exclusively formula feed
6. Have sufficient command of Tagalog or English language to complete the informed consent and other study documents
7. Are willing and able to fulfill the requirements of the study protocol
8. Have reached the legal age of consent in the Philippines
9. Able to be contacted by telephone throughout the study

Exclusion Criteria:

1. Infants who are receiving any amount of supplemental human milk
2. Family history of siblings with documented cow's milk protein intolerance/allergy
3. Conditions requiring infant feedings other than those specified in the protocol

Ages: 21 Days to 35 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2015-04; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Infant Gastrointestinal Symptom Questionnaire Composite Index Score | 6 weeks

SECONDARY OUTCOMES:
Formula Intake volume | 6 weeks
Stool Consistency Score | 6 weeks
Infant Toddler Quality of Life Profile | 6 weeks
Baby Eating Behaviour Questionnaire Profile | 6 weeks
Infant Characteristics Questionnaire (ICQ) Profile | 6 weeks

OTHER OUTCOMES:
Clinician-reported GI Adverse Event Profile | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Elvira M Estorninos, MD, Principal Investigator — Asian Hospital and Medical Center
Locations (1):
- Asian Hospital and Medical Center, Alabang, Muntinlupa City, Philippines

REFERENCES:
- [Derived] Volger S, Estorninos EM, Capeding MR, Lebumfacil J, Radler DR, Scott Parrott J, Rothpletz-Puglia P. Health-related quality of life, temperament, and eating behavior among formula-fed infants in the Philippines: a pilot study. Health Qual Life Outcomes. 2018 Jun 8;16(1):121. doi: 10.1186/s12955-018-0944-5. PMID 29884187